CLINICAL TRIAL: NCT02004054
Title: Interest of Dynamic Measures of the Pupil in Optic Neuritis
Acronym: PCT-NORB
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: SC_CLL_2012-8; 2012-A01260-43 (Other: ID RCB)
Record Dates: First submitted 2013-11-29; First posted 2013-12-06 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Optic Neuritis
Keywords: multiple sclerosis; diameter pupil
MeSH Terms: conditions — Optic Neuritis; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- optic neurotis: measure of pupil diameter
  Interventions: Other: measure of pupil diameter

INTERVENTIONS:
Other: measure of pupil diameter — The measure will use infra-red cameras

SUMMARY:
The investigators' hypothesis is that measuring the PCTdynamics would be an easy and reliable symptom to evaluate in pathologies affecting the optic nerve

DETAILED DESCRIPTION:
Physiopathologic study aiming to assess the interest of measuring the lenght of pupil cycle in the dynamic study of the pupillary light reflex.

ELIGIBILITY:
Inclusion Criteria:

* patients with unilateral optic neuritis or with multiple sclerosis and an optic neuritis in the previous 5 years

Exclusion Criteria:

* previous history of ophthalmic and neurologic pathology
* anisocoria
* minor
* Patient with a measure of legal protection
* Pregnancy
* patient opposition to participation in the study
* no affiliation to social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with unilateral optic neuritis or with multiple sclerosis and an optic neuritis in the previous 5 years
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Comparison between the PCT frequency of the eye affected by optic neuritis and a sane eye | after 1h

CONTACTS AND LOCATIONS:
Overall Officials: Cédric Lamirel, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France